CLINICAL TRIAL: NCT05076526
Title: Randomized Controlled Trial Comparing Cellular Matrix Combination of Platelet Rich Plasma With Hyaluronic Acid (CM-PRP-HA) Versus Hyaluronic Acid in Knee Osteoarthritis
Brief Title: PRP-HA Versus HA in Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Kenon Chua Ser, Orthopaedic Surgery Registrar, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: In progress
Record Dates: First submitted 2021-07-01; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Platelet-rich plasma; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-blinded randomised controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA (Active Comparator): Patients will receive 2 intra-articular injections of 2mL Synolis VA (20 mg/mL HA and 40 mg/mL sorbitol), with an interval of 1 month between both injections.
  Interventions: Biological: Hyaluronic acid (Synolis VA)
- PRP-HA (Experimental): Patients will receive 2 intra-articular injections of 5mL CM-PRP-HA combination (3mL of autologous PRP, 2mL of 16mg/mL HA), with an interval of 1 month between both injections.
  Interventions: Biological: Cellular Matrix platelet-rich-plasma with hyaluronic acid (CM PRP-HA)

INTERVENTIONS:
Biological: Hyaluronic acid (Synolis VA) — Synolis VA harbours the following characteristics:
  * NaHA (Sodium hyaluronate): 20mg/mL, biofermantative and pharmaceutical grade origin.
  * Sorbitol: 40mg/mL
  * Molecular weight of 2MDa, sterilized in moist heat
  Arms: HA
Biological: Cellular Matrix platelet-rich-plasma with hyaluronic acid (CM PRP-HA) — The CM-PRP-HA tube is under vacuum containing the following:
  * 2mL of hyaluronic acid gel in phosphate buffer (Sodium chloride, Dipotassium hydrogenphosphate, Potassium dihydrogenphosphate, Potassium chloride and water for injection). Not crosslinked Hyaluronic Acid (40mg per tube) is obtained from fermentation
  * 3g of inert cell-selector gel
  * 0.6mL of anticoagulant (sodium citrate 4%)
  Arms: PRP-HA

SUMMARY:
Osteoarthritis (OA) is a prevalent chronic condition which most commonly affects the knee. The pathogenesis of OA involves initial mechanical stress resulting in cartilage lesions, leading to inflammatory processes causing joint degradation. Numerous pharmacological and non-pharmacological therapies have been employed, including hyaluronic acid (HA) supplementations to alleviate the joint damage from mechanical load by acting as a shock absorber which provides lubrication, and intra-articular corticosteroid injections to reduce inflammation. However, HA is unable to facilitate cartilage regeneration and corticosteroids has numerous undesirable side effects which render them unsustainable treatment options.

Recently, many studies worldwide have demonstrated that platelet-rich-plasma (PRP) stimulates cartilage repair by actively secreting growth factors which activate cell proliferation and differentiation thereby promoting tissue regeneration. However, there has been varying results across various RCTs due to the heterogeneity of studies, with inconclusive recommendations on the treatment regimen for PRP-HA. Currently, PRP treatment is also not formally recognized as a treatment modality for knee OA in many countries, including Singapore.

This randomised controlled trial aims to compare the efficacy of Cellular Matrix (CM) PRP-HA versus HA (Synolis VA) intra-articular injections in knee OA through quantifying the improvement in long-term treatment outcomes such as pain, stiffness, and functional impairment, potentially improving the quality of life for many patients with knee OA.

DETAILED DESCRIPTION:
In vitro experimentations have also established the efficacy of PRP, where chondrocytes stimulated with PRP has shown to increase proteoglycan and collagen synthesis which bears similar biochemical qualities to that of hyaline cartilage. PRP has also shown to provide more critical growth factors (including PDGF, TGF-beta, IGF, EGF, VEGF, FGF) than conventional culture media, increasing the synthesis of major cellular proteins and collagen in the extracellular component of intervertebral disc cells, potentially enhancing the functional properties of joint cartilages.

Presently, cellular matrix (CM) remains as the only device which allows for the combination of PRP and HA to be delivered to patients within a single intra-articular injection. However, there are insufficient large-scale studies to reliably evaluate the efficacy of PRP-HA on knee OA and formulate a universal recommendation on its treatment regimen. There are also no RCTs conducted on our local population to explore the effects of CM-PRP-HA on knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 30 years and above
* Radiographical diagnosis of knee OA - ie narrowing of joint space, presence of osteophytes, possible sclerosis and subchondral cysts
* History of chronic pain in knee or knee swelling for at least 3 months
* Ability of patients to provide informed consent

Exclusion Criteria:

* Concurrent complementary and alternative medicine (CAM) treatments e.g. acupuncture
* Inflammatory diseases / infection / fracture / trauma
* Malignancies
* Pregnant or lactating females
* Consistent use of NSAIDs within 48 hours of procedure
* Corticosteroid injection at treatment site within 1 month
* Systemic use of corticosteroids within 2 weeks
* Tobacco use
* (For patients receiving PRP-HA injection only): Hemoglobin <10 g/dL and platelets <150,000/mm3

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Baseline
  WOMAC score comprises pain score, stiffness score and functional impairment score. Pain scores range from 0 to 20, stiffness scores range from 0 to 8, functional impairment scores range from 0 to 68. Total WOMAC score, which is an addition of the above 3 components, range from 0 to 96. Higher scores indicate worse outcomes
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score from baseline at 1 month | 1 month after last injection
  WOMAC score comprises pain score, stiffness score and functional impairment score. Pain scores range from 0 to 20, stiffness scores range from 0 to 8, functional impairment scores range from 0 to 68. Total WOMAC score, which is an addition of the above 3 components, range from 0 to 96. Higher scores indicate worse outcomes
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score from baseline at 3 months | 3 months after last injection
  WOMAC score comprises pain score, stiffness score and functional impairment score. Pain scores range from 0 to 20, stiffness scores range from 0 to 8, functional impairment scores range from 0 to 68. Total WOMAC score, which is an addition of the above 3 components, range from 0 to 96. Higher scores indicate worse outcomes
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score from baseline at 6 months | 6 months after last injection
  WOMAC score comprises pain score, stiffness score and functional impairment score. Pain scores range from 0 to 20, stiffness scores range from 0 to 8, functional impairment scores range from 0 to 68. Total WOMAC score, which is an addition of the above 3 components, range from 0 to 96. Higher scores indicate worse outcomes

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be made available